CLINICAL TRIAL: NCT06425081
Title: Investigating the Impact of Humiome B2 (Colon Delivered Riboflavin) and Riboflavin-overproducer Probiotic Strain Limosilactobacillus Reuteri AMBV339 on Intestinal and Vaginal Microbiome and Health (The VIAB2L Project)
Brief Title: Investigating the Impact of Humiome B2 (Colon Delivered Riboflavin) and Riboflavin-overproducer Probiotic Strain Limosilactobacillus Reuteri AMBV339 on Intestinal and Vaginal Microbiome and Health of Healthy Adult Women (The VIAB2L Project)
Acronym: VIAB2L
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: 2023-07-14-VIAB
Record Dates: First submitted 2024-05-08; First posted 2024-05-22 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2024-09

CONDITIONS: Microbial Colonization
Keywords: Probiotic; vitamin; Riboflavin; Vitamin B2; lactobacillus; microbiome; gut microbiome; vaginal microbiome; women's health; gut health
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomized and placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- L. reuteri AMBV339 (Active Comparator): Probiotic strain, 1B AFU (per day for 28 days in capsule format)
  Interventions: Dietary Supplement: Limosilactobacillus reuteri AMBV339
- Humiome B2 (Active Comparator): 73 mg colon delivered riboflavin containing 10 mg pure riboflavin (per day for 28 days in capsule format)
  Interventions: Dietary Supplement: Humiome B2
- Combination arm (Active Comparator): Probiotic strain, 1B AFU + 73 mg colon delivered riboflavin containing 10 mg pure riboflavin (per day for 28 days in capsule format)
  Interventions: Dietary Supplement: Limosilactobacillus reuteri AMBV339 + Humiome B2
- Placebo (Placebo Comparator): Microcrystalline cellulose (per day for 28 days in capsule format)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Limosilactobacillus reuteri AMBV339 — Limosilactobacillus reuteri AMBV339 is a probiotic strain
  Arms: L. reuteri AMBV339
Dietary Supplement: Humiome B2 — Colon-delivered Riboflavin
  Arms: Humiome B2
Dietary Supplement: Limosilactobacillus reuteri AMBV339 + Humiome B2 — Combination of supplements used in arm 1 and 2
  Arms: Combination arm
Dietary Supplement: Placebo — Microcrystalline cellulose
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if the probiotic strain Limosilactobacillus reuteri AMBV339 or colon-delivered riboflavin or their combination can change the gut and vaginal microbiome and metabolomics. It will also learn about the safety of the investigational product. The main questions it aims to answer are:

Do the probiotic strain Limosilactobacillus reuteri AMBV339 or colon-delivered riboflavin or their combination modify gut microbiome? Do the probiotic strain Limosilactobacillus reuteri AMBV339 or colon-delivered riboflavin or their combination modify gut microbiome?

Researchers will compare the probiotic strain Limosilactobacillus reuteri AMBV339 or colon-delivered riboflavin or their combination to a placebo (a look-alike substance that contains no drug) to see if they can change gut and vaginal microbiome. Intervention period is 28 days.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn if the probiotic strain Limosilactobacillus reuteri AMBV339 or colon-delivered riboflavin or their combination can change the gut and vaginal microbiome and metabolomics. It will also learn about the safety of the investigational product. Participants are healthy adult females of reproductive age and will take the investigational products for 28 days. There will be several non-invasive measurements, including but not limited to gut microbiome measured in faecal samples and vaginal microbiome measured in vaginal samples. They will fill some questionnaires about their general health.

The investigational product is a probiotic strain (1 billion AFU), colon-delivered riboflavin,(10mg) and their combination.

Participants will:

Take the probiotic strain Limosilactobacillus reuteri AMBV339 or colon-delivered riboflavin or their combination or a placebo every day for 28 days.

Visit the clinic once every 2 weeks for checkups and tests. Keep a diary of their bowel habits and provide fecal and vaginal sample at visits.

ELIGIBILITY:
Inclusion Criteria:

* Women of reproductive age (appr. 18-45 years old)
* Women of self-reported good general health
* Living in Flanders and speaking Dutch
* Using a combination contraceptive pill (without stop week) during the study and preferably at least three months before the study OR having a hormonal intrauterine device during the study and preferably at least three months before the study
* Subjects willing and able to give written informed consent and to understand, to participate and to comply with the clinical study requirements.

Exclusion Criteria:

* Current pregnancy or breastfeeding
* Antibiotic/antimycotic use during the last three months before the study
* Use of group B vitamin supplements or vitamin C during the study (record vitamin use via questionnaires)
* Ketogenic diet during the study and during the last two weeks before the study
* Oral and vaginal probiotic, prebiotic, and postbiotic and synbiotic supplementation during the study or recent use during the last two weeks before the study
* Vaginal douching during the study
* Presence of general infection
* Having a reproductive disorder or current vaginal infection or vaginal symptoms (VVC, BV, AV, etc.)
* Having a gastro-intestinal disorder or current GIT infections or gastrointestinal disorders (Crohn, IBS, IBD, etc.)
* Having any other medical condition that gives rise to exclusion from the study according to the responsible clinician/principal investigator of the study
* Participation in another clinical trial

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 185 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Microbiome change in GUT | day 0 - day 28
  1. To investigate if daily supplementation (for 28 days) with either Humiome B2 or Limosilactobacillus reuteri AMBV339 or their combination modulate the microbiome composition (relative abundance of different taxa) in the gastrointestinal tract (GIT). Comparisons will be made between the active groups and with placebo.

SECONDARY OUTCOMES:
Microbiome change in vagina | day 0 - day 28
  To investigate if daily supplementation (for 28 days) with either Humiome B2 or L. reuteri AMBV339 or their combination modulate the microbiome composition (relative abundance of different taxa) in the vagina. Comparisons will be made between the active groups and with placebo.
Gut microbiome diversity | day 0 - day 28
  2. To investigate if daily supplementation (for 28 days) with either Humiome B2 or L. reuteri AMBV339 or their combination modulate the microbiome diversity in the GIT. Comparisons will be made between the active groups and with placebo.
Vaginal microbiome diversity | day 0 - day 28
  To investigate if daily supplementation (for 28 days) with either Humiome B2 or L. reuteri AMBV339 or their combination modulate the microbiome diversity in the vagina. Comparisons will be made between the active groups and with placebo.
Keystone bacterial taxa in gut | day 0 - day 28
  To investigate if daily supplementation (for 28 days) with either Humiome B2 or L. reuteri AMBV339 or their combination modulate the relative abundance levels of keystone taxa in the GIT. Comparisons will be made between the active groups and with placebo.
Keystone bacterial taxa in vagina | day 0 - day 28
  To investigate if daily supplementation (for 28 days) with either Humiome B2 or L. reuteri AMBV339 or their combination modulate the relative abundance levels of keystone taxa in the vagina. Comparisons will be made between the active groups and with placebo.
Presence of L. reuteri AMBV339 in gut | day 0 - day 28
  To investigate the effect of daily supplementation (for 28 days) with either L. reuteri AMBV339 or its combination with Humiome B2 on the presence, persistence and/or engraftment of L. reuteri AMBV339 in the GIT during the intervention and 1 week after the end of supplementation. Comparisons will be made between the active groups and with placebo.
Presence of L. reuteri AMBV339 in vagina | day 0 - day 28
  To investigate the effect of daily supplementation (for 28 days) with either L. reuteri AMBV339 or its combination with Humiome B2 on the presence, persistence and/or engraftment of L. reuteri AMBV339 in the vagina during the intervention and 1 week after the end of supplementation. Comparisons will be made between the active groups and with placebo.
co-occurrence patterns of different bacterial taxa in the Gut microbiome | day 0 - day 28
  To investigate the effect of daily supplementation (for 28 days) with either Humiome B2 or L. reuteri AMBV339 or their combination on co-occurrence patterns of different bacterial taxa in the GIT, with particular attention to the possible role of riboflavin as an extracellular electron transfer molecule. Comparisons will be made between the active groups and with placebo.
co-occurrence patterns of different bacterial taxa in the vaginal microbiome | day 0 - day 28
  To investigate the effect of daily supplementation (for 28 days) with either Humiome B2 or L. reuteri AMBV339 or their combination on co-occurrence patterns of different bacterial taxa in the vagina, with particular attention to the possible role of riboflavin as an extracellular electron transfer molecule. Comparisons will be made between the active groups and with placebo.
Gut metabolomic profile | day 0 - day 28
  To investigate if daily supplementation (for 28 days) with either Humiome B2 or L. reuteri AMBV339 or their combination modulate the metabolomic profile in the GIT. Comparisons will be made between the active groups and with placebo.
Vaginal metabolomic profile | day 0 - day 28
  To investigate if daily supplementation (for 28 days) with either Humiome B2 or L. reuteri AMBV339 or their combination modulate the metabolomic profile in the vagina. Comparisons will be made between the active groups and with placebo.
levels of riboflavin in the gut | day 0 - day 28
  To investigate the effect of daily supplementation (for 28 days) with either Humiome B2 or L. reuteri AMBV339 or their combination on the levels of riboflavin in the GIT. Comparisons will be made between the active groups and with placebo.
levels of riboflavin in vagina | day 0 - day 28
  To investigate the effect of daily supplementation (for 28 days) with either Humiome B2 or L. reuteri AMBV339 or their combination for 28 days on the levels of riboflavin in the vagina. Comparisons will be made between the active groups and with placebo.
systemic levels of riboflavin (in blood) | day 0 - day 28
  To investigate the effect of 28 days of supplementation with either Humiome B2 or L. reuteri AMBV339 or their combination on the systemic levels of riboflavin (in blood). Comparisons will be made between the active groups and with placebo.
Short chain Fatty Acid (SCFA) levels in gut | day 0 - day 28
  To investigate the effect of daily supplementation (for 28 days) with either Humiome B2 or L. reuteri AMBV339 or their combination on the levels of short-chain fatty acids (SCFAs) and related metabolites in the GIT. Comparisons will be made between the active groups and with placebo.

OTHER OUTCOMES:
Excreted levels of riboflavin (in urine) | day 0 - day 28
  To investigate the effect of daily supplementation (for 28 days) with either Humiome B2 or L. reuteri AMBV339 or their combination on the excreted levels of riboflavin (in urine). Comparisons will be made between the active groups and with placebo.
Immune markers | day 0 - day 28
  To investigate the effect of 28 days of supplementation with either Humiome B2 or L. reuteri AMBV339 or their combination on key anti-inflammatory and cytokine markers in the vagina , assessed by ELISA (e.g., beta-defensin-1 and secretory IgA as well as a broad panel of protein biomarkers). Comparisons will be made between the active groups and with placebo.
General GIT health | day 0 - day 28
  To investigate the effect of daily supplementation (for 28 days) with either Humiome B2 or L. reuteri AMBV339 or their combination on GIT health will be measured using the GSRS questionnaire. Comparisons will be made between the active groups and with placebo.
General Vaginal health | day 0 - day 28
  To investigate the effect of daily supplementation (for 28 days) with either Humiome B2 or L. reuteri AMBV339 or their combination on general Vaginal health will measured using a Ph meter. Comparisons will be made between the active groups and with placebo.
General host health: Body temperature | day 0 - day 28
  To investigate the effect of daily supplementation (for 28 days) with either Humiome B2 or L. reuteri AMBV339 or their combination on host Body temperature using a thermometer. Comparisons will be made between the active groups and with placebo.
General host health: Pulse rate | day 0 - day 28
  To investigate the effect of daily supplementation (for 28 days) with either Humiome B2 or L. reuteri AMBV339 or their combination on host Pulse rate using a pulse rate monitor. Comparisons will be made between the active groups and with placebo.
General host health: Respiration rate | day 0 - day 28
  To investigate the effect of daily supplementation (for 28 days) with either Humiome B2 or L. reuteri AMBV339 or their combination on host Respiration rate by counting the number of chest rises per minute in rest mode. Comparisons will be made between the active groups and with placebo.
General host health: Blood pressure | day 0 - day 28
  To investigate the effect of daily supplementation (for 28 days) with either Humiome B2 or L. reuteri AMBV339 or their combination on host Blood pressure sphygmomanometer. Comparisons will be made between the active groups and with placebo.
User satisfaction of investigational product | day 0 - day 28
  To investigate the effect of daily supplementation (for 28 days) with either Humiome B2 or L. reuteri AMBV339 or their combination on user satisfaction levels based on a simple questionnaire of 10 point scale of how they felt before and after intervention (0 being the lowest point and 10 being the highest point). Comparisons will be made between the active groups and with placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Verhoeven, Dr, Principal Investigator — University of Antwerp Department of Family Medicine and Population Health; Sarah Lebeer, Dr, Principal Investigator — University of Antwerp Department of Bioscience Engineering
Locations (1):
- Lab of Applied Microbiology and Biotechnology, University of Antwerp, Antwerp, Antwerp, Belgium